CLINICAL TRIAL: NCT03778333
Title: Mesenchymal Stem Cells for Progressive Multiple Sclerosis_Sweden
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Lou Brundin, MD, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC-progressive MS
Record Dates: First submitted 2015-01-14; First posted 2018-12-19 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Autologous Mesenchymal Stem Cells; Multiple Sclerosis
Keywords: Mesenchymal Stem Cells; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Open-label phase 1, single-center, pre-post comparison study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label single arm study (Experimental): All patients will be treated with 1 single dose of IV infusion of autologous bone-marrow derived mesenchymal stem cells (1-2 million cells/kg body weight) and their therapeutic response will be followed over 48 weeks.
  Interventions: Biological: Autologous mesenchymal stem cells

INTERVENTIONS:
Biological: Autologous mesenchymal stem cells — IV therapy with autologous bone-marrow derived mesenchymal stem cells

SUMMARY:
To assess the safety of a single dose of IV infusion of bone-marrow derived autologous Mesenchymal Stem Cells (MSCs) in Multiple Sclerosis (MS) with progressive disease status.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MS

   1. Active relapsing remitting MS (RRMS) as evidenced by presence of ≥ 1 clinically documented relapse in the past 12 months or ≥2 clinically documented relapses in the last 24 months.
   2. Secondary progressive MS with clinical progression as evidenced by an increase of 1 EDSS point (or 0,5 p if EDSS ≥ 5 at time for study start) in the last year or evidenced by ≥1 relapse or ≥ GEL at MRI performed within the last year.
   3. Primary progressive MS with clinical progression as evidenced by an increase of 1 EDSS point (or 0,5 p if EDSS ≥ 5 at time for study start) in the last year.
2. Age_ 18-65 years
3. Disease duration: 2-20 years
4. EDSS 3,0-7,0

Exclusion Criteria:

1. Subtype of MS not fulfilling inclusion criteria
2. Treatment with any immunosuppressive therapy, including natalizumab and fingolimod, within the 3 months prior to randomization
3. Treatment with interferon-beta or glatiramer acetate within the 30 days prior to randomization
4. Treatment with corticosteroids within the 30 days prior to randomization
5. Relapse occurred during the 60 days prior to randomization
6. Previous history of a malignancy other than basal cell carcinoma of the skin or carcinoma in situ that has been in remission for more than one year
7. Severely limited life expectancy by another co-morbid illness
8. Active or chronic severe infection.
9. History of previous diagnosis of myelodysplasia or previous hematologic disease or current clinically relevant abnormalities of white blood cell counts
10. Pregnancy or risk or pregnancy (this includes patients that are unwilling to practice active contraception during the duration of the study)
11. eGFR < 60 mL/min/1.73m2 or known renal failure or inability to undergo MRI examination.
12. Inability to give written informed consent in accordance with research ethics board guidelines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
To evaluate number of participants with an adverse event related to the treatment. | 48 weeks
  Adverse events is defined as any untoward or undesirable medical occurence in the form of signs, symptoms, abnormal findings or diseases that emerge during the study period, regardless of causal relationship to the study drug.
To evaluate effects on MS disease activity measured by cumulative number of MRI T2 lesions. | 48 weeks
  Brain MRI examination

SECONDARY OUTCOMES:
To evaluate effects on MS disease activity measured by change in EDSS (expanded disability status scale). | 48 weeks
  EDSS assessed by neurologist.
To evaluate effect on peripheral blood immune cell populations. | 24 weeks
  Peripheral blood samples.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Karolinska Institute, Karolinska University Hospital Solna, Stockholm
  - Karolinska Institute, Karolinska University Hospital, Stockholm